CLINICAL TRIAL: NCT07059338
Title: Trastuzumab in Combination With Cetuximab and Irinotecan for the Treatment of HER2-Positive Metastatic Colorectal Cancer：A Phase II, Open-Label Trial
Brief Title: Dual EGFR/HER2 Blockade Combined With Irinotecan for the Treatment of HER2-Positive Metastatic Colorectal Cancer
Acronym: HERBIC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-160
Record Dates: First submitted 2025-06-05; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: HER2 Positive; Colorectal Cancer (CRC)
Keywords: colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab +Cetuximab β+Irinotecan (Experimental): Treatment regimen: All agents will be administered via intravenous infusion, consisting of trastuzumab (4 mg/kg every 2 weeks), cetuximab beta (500 mg/m² every 2 weeks) in combination with irinotecan (180 mg/m² every 2 weeks). Comprehensive radiological and laboratory assessments will be conducted after every 4 treatment cycles (8 weeks).
  Interventions: Drug: Trastuzumab +Cetuximab β+Irinotecan

INTERVENTIONS:
Drug: Trastuzumab +Cetuximab β+Irinotecan — Trastuzumab 4 mg/kg , Cetuximab β: 500 mg/m² ,Irinotecan 180 mg/m², repeat once every 2 weeks
  Other Names: HER2 and EGFR dual-targeted therapy combined with irinotecan

SUMMARY:
In colorectal cancer (CRC), HER2 has emerged as a critically targeted biomarker in recent years. Although multiple clinical trials have demonstrated the potential of HER2-targeted therapies in HER2-positive (overexpressed/amplified) metastatic CRC (mCRC), the duration of treatment response remains short with rapid disease progression. This underscores the urgent need to develop novel therapeutic strategies for HER2-positive mCRC. The EGFR pathway is constitutively activated in CRC and mediates resistance to HER2-targeted therapies through the formation of EGFR-HER2 heterodimers. Notably, EGFR-targeting antibodies combined with irinotecan can reverse irinotecan chemoresistance. Building upon these mechanisms, this study proposes to evaluate the combination of trastuzumab (anti-HER2), cetuximab beta (anti-EGFR), and irinotecan in chemotherapy-refractory HER2-positive mCRC.

DETAILED DESCRIPTION:
In colorectal cancer (CRC), HER2 has emerged as a significant therapeutic target, with clinical studies demonstrating promising yet transient responses to HER2-targeted therapies in HER2-positive (overexpressed/amplified) advanced cases, highlighting the need for improved strategies. Mechanistically, in the 65-75% of CRCs exhibiting EGFR overexpression, HER2 promotes heterodimerization with EGFR, impairing internalization of HER2-targeted ADCs and reducing drug uptake. Preclinical evidence suggests EGFR monoclonal antibodies (cetuximab/panitumumab) may overcome this limitation by inducing EGFR internalization and enhancing HER2-targeted drug efficacy. However, HER2-positive advanced CRC lacks validated predictive biomarkers and thorough translational research. Our study will clinically evaluate trastuzumab plus cetuximab and irinotecan in this population, while performing longitudinal biomarker analyses of paired blood and tumor samples to identify response predictors, elucidate resistance mechanisms, and optimize this promising therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent must be obtained voluntarily from the subject prior to performing any study-related procedures (non-routine care), in accordance with regulatory and institutional guidelines.
* 18 to 75 years of age, inclusive.
* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum with evidence of distant metastasis.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* HER2-positive tumor with wild-type KRAS, NRAS, and BRAF genes confirmed by testing at any time prior to screening. HER2 positivity is defined as: Immunohistochemistry (IHC) showing HER2 3+ staining in >50% of tumor cells; or HER2 2+ by IHC with positive fluorescence in situ hybridization (FISH): HER2/CEP17 ratio ≥2.0 in >50% of tumor cells; or Next-generation sequencing (NGS) of tissue or circulating tumor DNA (ctDNA) demonstrating HER2 copy number ≥6.
* Adequate organ function as evidenced by:

Absolute neutrophil count ≥1.5×10^9/L Platelet count ≥75×10^9/L Serum total bilirubin ≤1.5×upper normal limit (UNL) Aspartate aminotransferase (AST) ≤2.5×UNL Alanine aminotransferase (ALT) ≤2.5×UNL Serum creatinine ≤1.5×UNL

* Disease progression after prior treatment with fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy, including: Subjects who received oxaliplatin in the adjuvant setting must have experienced disease progression within 6 months after completing adjuvant therapy.Patients who decline standard therapy due to intolerable toxicity are eligible.
* Presence of at least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Willing and able to comply with the study protocol and visit schedule

Exclusion Criteria:

* Known KRAS, NRAS, or BRAF mutations detected by ctDNA testing prior to enrollment; or tumors with mismatch repair deficiency (dMMR) or high microsatellite instability (MSI-H).
* Concurrent intestinal obstruction, active bleeding, or perforation requiring emergency surgery.
* Major surgery (e.g., laparotomy, thoracotomy, or organ resection via laparoscopy) or significant trauma within 4 weeks prior to study entry (surgical incision must be fully healed before enrollment).
* Active coronary artery disease within 12 months before screening, including severe/unstable angina, newly diagnosed angina, or myocardial infarction.
* History of thrombosis or embolism within 6 months, including cerebrovascular accident (transient ischemic attack included), pulmonary embolism, or deep vein thrombosis.
* Congestive heart failure classified as New York Heart Association (NYHA) Class II or higher.
* HIV infection or AIDS; untreated active hepatitis (HBV-DNA ≥500 IU/mL for hepatitis B; detectable HCV-RNA for hepatitis C); or HBV/HCV co-infection.
* Interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, acute pneumonia).
* Persistent ≥Grade 2 toxicities (per CTCAE v5.0) from prior therapies (excluding peripheral neuropathy, anemia, alopecia, or skin hyperpigmentation).
* Known or suspected hypersensitivity to any study drugs.
* Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-11 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free-survival rates | 2 years
  Progression-free survival defined as the time from randomization to documented disease progression according to RECIST or death from any cause. We computed the 6-month PFS rate based on the available follow-up data.

SECONDARY OUTCOMES:
Objective response rate | 2 years
  defined as the percentage of patients with complete or partial response according to RECIST
Disease control rate | 2 years
  defined as the percentage of patients with CR + PR + SD according to RECIST
overall survival | 3 years
  defined as the time from randomization to death from any cause
Incidence of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 years
  Percentage of patients, experiencing a specific adverse event, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during the induction and the maintenance phases of treatment.

OTHER OUTCOMES:
Treatment-emergent genetic variants analysis by ctDNA sequencing | 2 years
  Longitudinal assessment of somatic mutation profiles in circulating tumor DNA (ctDNA) using next-generation sequencing (NGS) to correlate genetic variants (e.g., HER2/EGFR/RAS pathway alterations) with objective response rate (ORR) per RECIST 1.1 criteria.
Baseline proteomic predictive biomarkers for treatment efficacy | 3 years
  Quantitative proteomic profiling of baseline plasma and tissue samples to identify predictive biomarkers correlated with therapeutic response.
Treatment-induced proteomic alterations | 3 years
  Quantitative proteomic analysis of plasma and tissue samples to detect therapy-mediated changes in protein expression and phosphorylation patterns.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No